CLINICAL TRIAL: NCT02935842
Title: Effectiveness of High-frequency Specific Speech Therapy on Verbal Fluency Decline and/ or Verbal Apraxia in Patients With Parkinson's Disease With and Without Deep Brain Stimulation (DBS) - a Randomized Controlled Single-blinded Trial
Brief Title: Evaluation of Intensive Language Therapy
Acronym: EILT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: EILT
Record Dates: First submitted 2016-08-18; First posted 2016-10-18 (Estimated); Results first posted 2020-06-02 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; Word Retrieval; Apraxia Symptoms; Dysarthria
MeSH Terms: conditions — Parkinson Disease; Dysarthria

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Specific SL-therapy for PD (with and without DBS) (Experimental): Rhythmic specific, intensive and high-frequency SL-therapy. Approx. 45 Min. per session, 3 times per week for 4 weeks
  Interventions: Other: Specific SL-therapy; Other: Rhythmic Balance-Movement Training (rBMT)
- rBMT for PD (with and without DBS) (Active Comparator): Rhythmic Balance-Movement Training (rBMT); approx. 30-45 Minutes per session, 3 times per week for 4 weeks
  Interventions: Other: Specific SL-therapy; Other: Rhythmic Balance-Movement Training (rBMT)
- PD (with and without DBS); no therapy (No Intervention): No further recruiting necessary, as data is already at hand via previous research projects.
- Healthy Controls; no therapy (No Intervention): No further recruiting necessary, as data is already at hand via previous research projects.

INTERVENTIONS:
Other: Specific SL-therapy — Provided by a professional speech-language therapist (SLT) on a one-to-one basis. In approx. 45 Minutes sessions, 3 times per week for 4 weeks in total.
  Other Names: Specific, intensive and high-frequency SL-therapy
  Arms: Specific SL-therapy for PD (with and without DBS); rBMT for PD (with and without DBS)
Other: Rhythmic Balance-Movement Training (rBMT) — Provided on a one-to-one basis. In approx. 30-45 Minutes sessions, 3 times per week for 4 weeks in total.
  Arms: Specific SL-therapy for PD (with and without DBS); rBMT for PD (with and without DBS)

SUMMARY:
Due to Parkinson's Disease (PD) speech and language (SL) deficits may occur. Further, the literature reports that PD patients, who have not undergone deep brain stimulation (DBS), have deficits regarding voice quality (e.g. loudness and intelligibility of their voice), while PD patients who have undergone DBS suffer from deficits in word retrieval and speech apraxia symptoms. To-date, therapeutic approaches focusing specifically on SL deficits observed in PD-DBS patients are yet to be developed and evaluated.

Therefore, this study investigates the short-and longterm effectiveness of specific and intensive, high-frequency speech-language therapy in terms of reducing SL-deficits compared to a nonspecific and non-verbal sham treatment (i.e. a rhythmic balance-movement training (rBMT)) as well as to a 'no-therapy' condition.

DETAILED DESCRIPTION:
In the course of Parkinson's disease (PD) speech and language (SL) deficits may often emerge. In addition, severe verbal fluency (VF) decline has been repeatedly observed in the context of deep brain stimulation (DBS) in PD. Interestingly, while PD non-DBS patients have deficits with respect to loudness and intelligibility of their voice, PD patients who have undergone DBS (PD-DBS) suffer rather from difficulties in semantic and phonemic word retrieval, and from speech apraxia symptoms.

However, to-date and to the best of our knowledge, therapeutic approaches focusing specifically on SL deficits observed in PD-DBS patients are yet to be developed and evaluated regarding their effectiveness. Thus, this study investigates the short-and longterm effectiveness of specific and intensive, high-frequency speech-language therapy in terms of reducing SL-deficits compared to a nonspecific and non-verbal sham treatment (i.e. a rhythmic balance-movement training (rBMT)) as well as to a 'no-therapy' condition.

ELIGIBILITY:
Inclusion Criteria for all groups:

* The patient is able to cooperate
* The patient has the mental competence to provide informed consent to participate in the study
* The patient speaks and understands German

Specific Inclusion Criteria for the DBS Group

* Fulfilling the above stated inclusion criteria as stated in a, b and c above
* The patient is responsive to Levodopa (L-DOPA)
* Having received or being scheduled for DBS

Exclusion Criteria:

* Severe psychiatric disease difficult to treat (compulsive disorder, depression, mania, psychosis, anxiety as outlined in International Classification of Diseases (ICD-10) (WHO 2015, current version).
* Patient with dementia (DMS-V, Mini-Mental-Status-Test (MMS) <24, Montreal Cognitive Assessment (MoCa) <21)
* Secondary Parkinsonism
* Age ≤18 years
* Pregnancy (early onset)
* Presence of a known disease other than PD that shortens the life expectancy
* Mental incompetence to provide informed consent to participate in the study
* Previous intracranial surgery
* Epilepsy
* Contraindications for DBS seen in MRI-scan (malignant tumour, severe microvascular disease)
* Insufficient skills of German language for participating in neuropsychological evaluations
* Sensory problems, severe enough to significantly interfere with neuropsychological assessment
* Alcohol and/or drug addiction

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2018-09-12 (Actual); Study Completion 2018-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Fuhr, Prof.Dr.med., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roesch AD, Gschwandtner U, Handabaka I, Meyer A, Taub E, Fuhr P. Effects of Rhythmic Interventions on Cognitive Abilities in Parkinson's Disease. Dement Geriatr Cogn Disord. 2021;50(4):372-386. doi: 10.1159/000519122. Epub 2021 Oct 28. PMID 34808624

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From May 2015 to February 2018, N=32 patients with idiopathic Parkinson's disease (PD) were recruited from the University Hospital Basel (Switzerland) and N=22 healthy controls (HC) were recruited from senior health centers or sports groups independent of the hospital.
Pre-assignment Details: Eligibility assessments were conducted by neurologists, neuropsychologists and speech-language therapists. Eligibility criteria led to 12 exclusions in the PD group and to 4 exclusions in the HC group.
  Therefore, final N count for the study were: N=20 PD patients and N=18 HC.
Groups:
- rSLT, Then no Therapy, Then rBMT: Specific, intensive and high-frequency speech-language-therapy (rSLT). Approx. 45 Min. per session, 3 times per week for 4 weeks
  Specific SL-therapy: Provided by a professional speech-language therapist (SLT) on a one-to-one basis. In approx. 45 Minutes sessions, 3 times per week for 4 weeks in total.
  Please note: this was a case-crossover study. Participants, who completed the above stated and described intervention, had then the opportunity to switch to the 'no therapy' group. After having completed the 6 months 'no therapy' period, the participant could enrol again into the 'rhythmic balance-movement training'' rBMT).
- rBMT, Then 'no Therapy', Then rSLT: Rhythmic Balance-Movement Training (rBMT); approx. 30-45 Minutes per session, 3 times per week for 4 weeks
  Rhythmic Balance-Movement Training (rBMT): Provided on a one-to-one basis. In approx. 30-45 Minutes sessions, 3 times per week for 4 weeks in total.
  Please note: this was a case-crossover study. Participants, who completed the above stated and described intervention, had then the opportunity to switch to the 'no therapy' group. After having completed the 6-months period as 'no therapy', the participant could switch to the 'rhythmic speech-language therapy' group (rSLT).
- No Therapy, Then rSLT, Then rBMT: "the 6-months-waiting list". Patients with Parkinson's disease (PD) who had to wait for/ or chose to receive treatments at a later time.
  Please note: this was a case-crossover study. After completing the 6-month waiting list (no therapy), participants had then the opportunity to switch to another study arm (being 'rhythmic speech-language therapy' (rSLT) or 'rhythmic balance-movement training' (rBMT). After having completed the second intervention program, the participant could enrol again into a study arm, which he/she has not been before (i.e. either 'rhythmic speech-language therapy' (rSLT) or 'rhythmic balance-movement training'' rBMT).
- Healthy Controls; no Therapy: Healthy Controls received no therapy.
Period: Testing and Therapy Period 1
Arm/Group | rSLT, Then no Therapy, Then rBMT | rBMT, Then 'no Therapy', Then rSLT | No Therapy, Then rSLT, Then rBMT | Healthy Controls; no Therapy
Started | 8 | 6 | 6 | 0 (Due to limited staff capacity, HC have only been included in the final tranche.)
Completed | 8 | 6 | 6 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Testing and Therapy Period 2
Arm/Group | rSLT, Then no Therapy, Then rBMT | rBMT, Then 'no Therapy', Then rSLT | No Therapy, Then rSLT, Then rBMT | Healthy Controls; no Therapy
Started | 8 | 6 | 6 | 0 (Due to limited staff capacity, HC have only been included in the final tranche.)
Completed | 6 | 6 | 6 | 0
Not Completed | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0
Period: Testing and Therapy Period 3
Arm/Group | rSLT, Then no Therapy, Then rBMT | rBMT, Then 'no Therapy', Then rSLT | No Therapy, Then rSLT, Then rBMT | Healthy Controls; no Therapy
Started | 6 | 6 | 6 | 18 (HC received no interventions. They have only been tested at BL, 4 Weeks and 6 Months.)
Completed | 3 | 2 | 1 | 17
Not Completed | 3 | 4 | 5 | 1
Not completed — Required other therapy (dysphagia) | 1 | 2 | 2 | 0
Not completed — Accident prior to treatment | 2 | 2 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Population: In this cross-over study, there were 20 PD patients and 18 healthy controls enrolled (HC final N=17, because on participant was lost to Follow-up).This baseline analysis gives all information per group, and PD patients could switch between the different groups (i.e. rSLT, rBMT, NT).
Groups:
- rSLT, Then no Therapy, Then rBMT: Specific, intensive and high-frequency SL-therapy. Approx. 45 Min. per session, 3 times per week for 4 weeks
  Specific SL-therapy: Provided by a professional speech-language therapist (SLT) on a one-to-one basis. In approx. 45 Minutes sessions, 3 times per week for 4 weeks in total.
  Then participants could be allocated to the no-therapy group, and after 6-month completion again into the rBMT intervention.
- rBMT, Then rSLT, Then no Therapy: Rhythmic Balance-Movement Training (rBMT); approx. 30-45 Minutes per session, 3 times per week for 4 weeks
  Rhythmic Balance-Movement Training (rBMT): Provided on a one-to-one basis. In approx. 30-45 Minutes sessions, 3 times per week for 4 weeks in total.
  Then participants could be enrolled in the rSLT group, and after 6-month completion again into the 'no-therapy' group.
- No Therapy, Then rSLT or rBMT, Then rBMT or rSLT: "the 6-months-waiting list". PD patients who had to wait for/ or chose to receive treatments at a later time.
  After 6-month completion, participants could enrol in the rSLT or the rBMT intervention program, and then upon 6-month completion again in the opposite intervention program, being rBMT or rSLT, respectively.
- Total: Total of all reporting groups
Arm/Group | rSLT, Then no Therapy, Then rBMT | rBMT, Then rSLT, Then no Therapy | No Therapy, Then rSLT or rBMT, Then rBMT or rSLT | Healthy Controls; no Therapy | Total
Number analyzed (Participants) | 8 | 6 | 6 | 17 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.4 (7.1) | 69.9 (6.7) | 65.1 (6.7) | 67.9 (5.2) | 68.9 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 2 | 10 | 18
  Male | 5 | 3 | 4 | 7 | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Switzerland | 8 | 6 | 6 | 17 | 37
Speech Velocity [Mean (Standard Deviation); unit: spoken syllables per second] | 5.3 (.6) | 5.3 (.6) | 4.9 (.4) | 2.3 (1.6) | 4.4 (1.4)
Speech Cadence [Mean (Standard Deviation); unit: Spoken syllables per inspiration] | 8.4 (3.5) | 9 (3.9) | 8.2 (.6) | 21.6 (.6) | 12.2 (7.4)
Gait velocity [Mean (Standard Deviation); unit: meters per second] | 1.3 (.4) | 1.2 (.4) | 1.2 (.3) | .8 (.08) | 1.2 (.4)
Gait Cadence [Mean (Standard Deviation); unit: steps per second] | 2.7 (.8) | 2.7 (.8) | 2.7 (.7) | 1.7 (.2) | 2.5 (.8)

OUTCOME MEASURES:

1. Primary Outcome: Velocity in Gait
Description: Gait Velocity: meters per second
Time Frame: At Baseline (BL), T1 after 4 weeks (4W-directly after intervention), T2 after 6 months (6M).
Measure: Mean (Standard Deviation); unit: meter per second
Groups:
- Specific SL-therapy for PD-DBS and Non-DBS: Specific, intensive and high-frequency SL-therapy. Approx. 45 Min. per session, 3 times per week for 4 weeks
  Specific SL-therapy: Provided by a professional speech-language therapist (SLT) on a one-to-one basis. In approx. 45 Minutes sessions, 3 times per week for 4 weeks in total.
- rBMT for PD-DBS and Non-DBS: Rhythmic Balance-Movement Training (rBMT); approx. 30-45 Minutes per session, 3 times per week for 4 weeks
  Rhythmic Balance-Movement Training (rBMT): Provided on a one-to-one basis. In approx. 30-45 Minutes sessions, 3 times per week for 4 weeks in total.
- PD-DBS/ Non-DBS; no Therapy: "the 6-months-waiting list". PD patients who had to wait for/ or chose to receive treatments at a later time.
Arm/Group | Specific SL-therapy for PD-DBS and Non-DBS | rBMT for PD-DBS and Non-DBS | PD-DBS/ Non-DBS; no Therapy | Healthy Controls; no Therapy
Number analyzed (Participants) | 16 | 10 | 18 | 17
meter per second
  Gait Velocity-4W (4Weeks) | 1.2 (.2) | 1.2 (.3) | 1.2 (.3) | .8 (.08)
  Gait Velocity-6M (6 Months) | 1.3 (.8) | 1.2 (.4) | 1.2 (.3) | .8 (.08)
Statistical Analysis 1: Comparison: Specific SL-therapy for PD-DBS and Non-DBS vs rBMT for PD-DBS and Non-DBS vs PD-DBS/ Non-DBS; no Therapy vs Healthy Controls; no Therapy; First Reliable Change (RC), Reliable Change Index (RCI) were calculated on every individual score. Further, ANOVAs and t-tests were administered in order to verify differences between groups or interventions. Significance levels were set at p < .05; Test type: Other; Reliable Change / Reliable Change Index according to Jacobson & Truax (1991). There, on the basis of every individual score, the change in performance (i.e. BL-4Weeks/ BL-6Months) has been calculated and is reported with level of significance as well as effect size
Statistical Analysis 2: Comparison: Specific SL-therapy for PD-DBS and Non-DBS vs rBMT for PD-DBS and Non-DBS vs PD-DBS/ Non-DBS; no Therapy vs Healthy Controls; no Therapy; Test type: Other; p = .05, ANOVA

2. Primary Outcome: Cadence in Gait
Description: 4-Weeks and 6-Months Follow-up. To measure rhythmicity in gait, participants walked 6 metres at their individual pace. They were timed and amount of steps were counted.
Time Frame: At Baseline (BL), T1 after 4 weeks (4W-directly after intervention), T2 after 6 months (6M).
Measure: Mean (Standard Deviation); unit: steps per second
Arm/Group | Specific SL-therapy for PD (With and Without DBS) | rBMT for PD (With and Without DBS) | PD (With and Without DBS); no Therapy | Healthy Controls; no Therapy
Number analyzed (Participants) | 16 | 10 | 18 | 17
steps per second
  Gait Cadence-4W | 2.5 (.3) | 2.5 (.6) | 2.7 (.7) | 1.7 (.2)
  Gait Cadence-6M | 2.8 (.8) | 2.7 (.8) | 2.7 (.7) | 1.7 (.2)

3. Primary Outcome: Speech Velocity
Description: Speech Velocity at 4 weeks and at 6 months
  To measure rhythmicity in speech, participants read a text aloud ('the north wind and the sun') and were recorded using an Olympus. According to these speech samples, the count of elicited syllables per second was calculated.
Time Frame: At Baseline (BL), T1 after 4 weeks (4W-directly after intervention), T2 after 6 months (6M).
Measure: Mean (Standard Deviation); unit: spoken syllables per second
Arm/Group | rSLT, Then no Therapy, Then rBMT | rBMT, Then rSLT, Then no Therapy | No Therapy, Then rSLT or rBMT, Then rBMT or rSLT | Healthy Controls; no Therapy
Number analyzed (Participants) | 16 | 10 | 18 | 17
spoken syllables per second
  Speech velocity 4W | 3.6 (.7) | 4.2 (.9) | 4.9 (.7) | 2.3 (.6)
  Speech velocity 6M | 3.8 (.8) | 4.8 (.9) | 4.9 (.6) | 2.3 (.6)

4. Primary Outcome: Speech Cadence
Description: Speech Cadence 4 Weeks and at 6 Months To measure rhythmicity in speech, participants' speech was recorded while reading a text aloud ('the north wind and the sun'). Elicited syllables per inspiration were analysed.
Time Frame: At Baseline (BL), T1 after 4 weeks (4W-directly after intervention), T2 after 6 months (6M).
Measure: Mean (Standard Deviation); unit: spoken syllables per inspiration
Arm/Group | rSLT, Then no Therapy, Then rBMT | rBMT, Then rSLT, Then no Therapy | No Therapy, Then rSLT or rBMT, Then rBMT or rSLT | Healthy Controls; no Therapy
Number analyzed (Participants) | 16 | 10 | 18 | 17
spoken syllables per inspiration
  Speech Cadence 4W | 15.6 (3.6) | 13.1 (4.7) | 10.9 (3.9) | 21.6 (6)
  Speech Cadence 6M | 13.3 (4.6) | 13.6 (4.7) | 10.5 (3.5) | 21.6 (6)

5. Secondary Outcome: Health Status (UPDRS)
Description: The complete questionnaire 'Unified Parkinson's Disease Rating Scale' (UPDRS) was filled out at BL and 6M.
  Scores may range from 0-4 per question. Final scores may add up to 199 points maximum. The higher the score, the worse disease severity/ degree of disability is.
Time Frame: At Baseline and 6 Months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Specific SL-therapy for PD-DBS and Non-DBS | rBMT for PD-DBS and Non-DBS | PD-DBS/ Non-DBS; no Therapy | Healthy Controls; no Therapy
Number analyzed (Participants) | 16 | 10 | 18 | 17
score on a scale
  UPDRS-BL | 38.6 (19.1) | 37.3 (20.6) | 42.8 (20.2) | 0 (0)
  UPDRS-6M | 35.6 (16.7) | 41.7 (19.1) | 37 (20.1) | 0 (0)
Statistical Analysis 1: Comparison: Specific SL-therapy for PD-DBS and Non-DBS vs rBMT for PD-DBS and Non-DBS vs PD-DBS/ Non-DBS; no Therapy vs Healthy Controls; no Therapy; Test type: Other; p = .05, ANOVA

6. Secondary Outcome: Neuropsychiatric Self-rating Questionnaires
Description: Self-rating questionnaires investigating depression using the Beck's Depression Inventory (BDI).
  This is a 21 question, multiple choice, self-report questionnaire. Minimum score is 0 and maximum scores is 63. The higher the score the more severe is the depression.
  Details:
  0-9: indicates minimal depression 10-18: indicates mild depression 19-29: indicates moderate depression 30-63: indicates severe depression.
Time Frame: At 4 Weeks and 6 Months
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Specific SL-therapy for PD-DBS and Non-DBS | rBMT for PD-DBS and Non-DBS | PD-DBS/ Non-DBS; no Therapy | Healthy Controls; no Therapy
Number analyzed (Participants) | 16 | 10 | 18 | 17
score
  BDI-4W | 8 (1.8) | 7.6 (2.1) | 7.1 (1.9) | 5.5 (2.2)
  BDI-6M | 7.4 (1.7) | 8.8 (1.6) | 8.3 (1.8) | 5.4 (2.2)

7. Secondary Outcome: Neuropsychological Standardised Test Battery
Description: Inhibition Control (Stroop), Visio-Construction (Mosaic), Flexibility (Trail Making Test), Episodic Memory (Basel Verbal Learning Test -long delayed free recall), Working Memory (backwards digit span task by Wechsler).
  Scores were standardized (z-scores) to a mean of 0 and standard deviation of 1. The Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean of a reference population. Negative numbers indicate values lower than the reference population and positive numbers indicate values higher than the reference population
Time Frame: At 4 Weeks and at 6 Months
Measure: Mean (Standard Deviation); unit: z-scores
Arm/Group | Specific SL-therapy for PD-DBS and Non-DBS | rBMT for PD-DBS and Non-DBS | PD-DBS/ Non-DBS; no Therapy | Healthy Controls; no Therapy
Number analyzed (Participants) | 16 | 10 | 18 | 17
z-scores
  Episodic Memory-4W | -.9 (1.7) | -.3 (1.2) | -.7 (.3) | -.4 (1.7)
  Episodic Memory-6M | -.7 (1.5) | -.6 (.8) | -.3 (1.1) | -.2 (1.1)
  Working Memory-4W | .6 (.8) | .2 (.9) | -.2 (.8) | .1 (1.7)
  Working Memory-6M | -.3 (1.1) | .13 (.9) | -.2 (.8) | -.5 (1.4)
  Visuo-Construction-4W | .4 (1.03) | .14 (1.1) | .4 (.9) | .4 (.8)
  Visa-Construction-6M | .03 (1) | .07 (.9) | .2 (.6) | .8 (1.05)
  Inhibition (Stroop)-4W | .6 (.8) | .8 (1.4) | .7 (.9) | .2 (1.3)
  Inhibition (Stroop)-6M | -.04 (.9) | .3 (.6) | .7 (.7) | .4 (.7)
  Flexibility (TMT)-4W | -.4 (.8) | -.6 (1.3) | -.8 (.3) | .2 (1.05)
  Flexibility (TMT)-6M | -.6 (1.02) | -1.2 (1.1) | -.3 (.8) | .8 (1.3)
Statistical Analysis 1: Comparison: Specific SL-therapy for PD-DBS and Non-DBS vs rBMT for PD-DBS and Non-DBS vs PD-DBS/ Non-DBS; no Therapy vs Healthy Controls; no Therapy; Test type: Other; p = .05, ANOVA

ADVERSE EVENTS:
Time Frame: Adverse Events were collected over the full length of the study for each participant. Beginning at the baseline measurement up to 1 year after completion.
Description: This cross-over study involved non-invasive intensive treatments (i.e. rhythmic speech therapy vs. rhythmic balance-mobility training).
Arm/Group | Specific SL-therapy for PD-DBS and Non-DBS | rBMT for PD-DBS and Non-DBS | PD-DBS/ Non-DBS; no Therapy | Healthy Controls; no Therapy
All-Cause Mortality (participants affected / at risk) | 0/20 | 1/20 | 0/20 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/18
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-09): https://cdn.clinicaltrials.gov/large-docs/42/NCT02935842/Prot_SAP_000.pdf